CLINICAL TRIAL: NCT05495139
Title: A Small-Sample-Size Clinical Study to Evaluate the Effectiveness and Safety of the Gastric Bypass Stent System in Treatment of Patients With Nonalcoholic Fatty Liver Disease.
Brief Title: Gastric Bypass Stent Small-Sample-Size Study For Nonalcoholic Fatty Liver Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Tangji Medical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZTJ03
Record Dates: First submitted 2022-08-07; First posted 2022-08-10 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single arm study, only investigational product (Experimental): To evaluate the preliminary effectiveness and safety of the Gastric Bypass Stent System in treating nonalcoholic fatty liver disease.
  Interventions: Device: Gastric Bypass Stent System in Treatment of Patients with Nonalcoholic Fatty Liver Disease

INTERVENTIONS:
Device: Gastric Bypass Stent System in Treatment of Patients with Nonalcoholic Fatty Liver Disease — This study includes 3 phases; screening period, procedural period, and a follow-up period. Following a 2-week screening period, subjects will be treated with the Gastric Bypass Stent System implanted under gastroscopy (Visit 2; Day 0). Following a 6-month treatment period, the device is removed, and subjects are followed for 6 months. In total subject participation will last for approximately 12 months.

SUMMARY:
Evaluate the preliminary effectiveness and safety of the Gastric Bypass Stent System in treating nonalcoholic fatty liver disease.

DETAILED DESCRIPTION:
The Gastric Bypass Stent System is intended to be used in Patients with Diagnosis of nonalcoholic fatty liver disease， Proton density fat fraction measured by magnetic resonance imaging (MRI-PDFF) ≥8%. In this pivotal, prospective, single-arm clinical investigation the Sponsor seeks to demonstrate the safety and performance of the Gastric Bypass Stent System in Treatment of Patients with Nonalcoholic Fatty Liver Disease

ELIGIBILITY:
Inclusion Criteria:

（ - ） Males or females with age between 18 and 65 years old;

（ - ） Diagnosis of nonalcoholic fatty liver disease;

（ - ） Proton density fat fraction measured by magnetic resonance imaging (MRI-PDFF) ≥8%;

（ - ） BMI≥24;

Patients who understand the objective of the study; voluntarily participate in the study and have signed the informed consent form; and are able and willing to comply with all requirements, including follow up and evaluations.

Exclusion Criteria:

（ - ） History of excessive alcohol consumption (alcohol consumption equivalent to ethanol > 30 g/d for males and > 20 g/d for females);

（ - ） End-stage liver disease (e.g. hepatic cirrhosis or hepatic cancer) or other conditions which may lead to fatty liver;

（ - ） Unable to cooperate to complete MR examination;

（ - ） Subjects who have used any nonsteroidal anti-inflammatory drug or corticosteroid in the past month;

（ - ） Patients with iron deficiency or iron deficiency anemia;

（ - ） ALT or AST increased to 8 × upper limit of normal (ULN), and bilirubin increased to 2×ULN;

（ - ） Patients with coagulation disorder or haemorrhagic diathesis (platelets <100×109/L);

（ - ） Patients with duodenal ulcer, or previous or existing pancreatitis;

（ - ） History of liver abscess;

（ - ） History of gallstones (symptomatic or presenting of any stone with a diameter greater than 20mm);

（ - ） Patients with gastrointestinal hemorrhage or potential hemorrhage;

（ - ） Gastrointestinal tract anomalies, such as gastrointestinal tract atresia or any or other conditions that would result in failed placement in the gastrointestinal tract;

（ - ） Patients with history of intestinal obstruction or related disease in the past year;

（ - ） Drug abusers or patients with uncontrollable psychiatric disorders;

（ - ） Patients with any contraindication to endoscopy based on the investigator's judgment;

（ - ） Pregnancy or lactating women;

（ - ） Patients who are participating in any other drug or medical device clinical study;

（ - ） Patients with any other conditions evaluated by the investigators as unsuitable for participating in the trial;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of MRI-PDFF | 24 weeks after device implantation procedure(Visit 7)
  Changes of MRI-PDFF at device retrieval

SECONDARY OUTCOMES:
Changes of MRI-PDFF | 12 weeks after device retrieval(Visit 8) and 24 weeks after device retrieval(Visit 9)
  Changes of MRI-PDFF at 12 and 24 weeks after device retrieval
Changes of liver stiffness measurement (LSM) | 24 weeks after the implantation procedure (Visit 7), and 12 weeks after device retrieval(Visit 8) and 24 weeks after device retrieval(Visit 9)
  Changes of liver stiffness measurement (LSM) at device retrieval, and 12 and 24 weeks after device retrieval
Changes of liver inflammation/injury indicators (ATL, ASL, GGT, ALP, TBil, and DBil) | 24 weeks after the implantation procedure (Visit 7), and 12 weeks after device retrieval(Visit 8) and 24 weeks after device retrieval(Visit 9)
  Changes of liver inflammation/injury indicators (ATL, ASL, GGT, ALP, TBil, and DBil) at device retrieval, and 12 and 24 weeks after device retrieval
Changes of blood glucose indicators (fasting insulin, fasting blood glucose, fasting C-peptide, and insulin resistance [e.g. HOMA-IR]) | 24 weeks after the implantation procedure (Visit 7), and 12 weeks after device retrieval(Visit 8) and 24 weeks after device retrieval(Visit 9)
  Changes of blood glucose indicators (fasting insulin, fasting blood glucose, fasting C-peptide, and insulin resistance [e.g. HOMA-IR]) at device retrieval, and 12 and 24 weeks after device retrieval
Changes of blood lipids indicators, including triglyceride, total cholesterol, low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), apolipoprotein A1, apolipoprotein B, apolipoprotein CIII, and lipoprotein (a) | 24 weeks after the implantation procedure (Visit 7), and 12 weeks after device retrieval(Visit 8) and 24 weeks after device retrieval(Visit 9)
  Changes of blood lipids indicators, including triglyceride, total cholesterol, low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), apolipoprotein A1, apolipoprotein B, apolipoprotein CIII, and lipoprotein (a), at device retrieval, and 12 and 24 weeks after device retrieval
Changes of hepatic fibrosis indicators (PIIINP, Fibro Test/Fibro Sure, ELF, and NFS) | 24 weeks after the implantation procedure (Visit 7), and 12 weeks after device retrieval(Visit 8) and 24 weeks after device retrieval(Visit 9)
  Changes of hepatic fibrosis indicators (PIIINP, Fibro Test/Fibro Sure, ELF, and NFS) at device retrieval, and 12 and 24 weeks after device retrieval
Percent changes of body weight and changes of BMI | 24 weeks after the implantation procedure (Visit 7), and 12 weeks after device retrieval(Visit 8) and 24 weeks after device retrieval(Visit 9)
  Percent changes of body weight and changes of BMI at device retrieval and 12 and 24 weeks after device retrieval
Histological changes | 24 weeks after the implantation procedure (Visit 7)
  Histological changes at device retrieval
Evaluation on the usability of the device | 4 weeks after the implantation procedure (Visit 4) 、12 weeks after the implantation procedure (Visit 5)and 18 weeks after the implantation procedure (Visit 6)
  Use abdominal X-ray evaluate Device implantation status

CONTACTS AND LOCATIONS:
Overall Officials: Lungen Lu, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Baiwen Li, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China